CLINICAL TRIAL: NCT00369577
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Single Dose Efficacy and Safety Study of StaccatoTM Loxapine for Inhalation in Schizophrenic Patients With Agitation.
Brief Title: Staccato Loxapine in Agitation (Proof of Concept)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-201; 004-201
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Agitation; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychomotor Agitation | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Placebo (Placebo Comparator): Inhaled Staccato Placebo, single dose
  Interventions: Drug: Inhaled Placebo
- Inhaled Loxapine 5 mg (Experimental): Inhaled Staccato Loxapine 5 mg, single dose
  Interventions: Drug: Inhaled Loxapine 5 mg
- Inhaled Loxapine 10 mg (Experimental): Inhaled Staccato Loxapine 10 mg, single dose
  Interventions: Drug: Inhaled Loxapine 10 mg

INTERVENTIONS:
Drug: Inhaled Placebo — Inhaled Placebo, single dose
  Other Names: Staccato Loxapine Placebo
  Arms: Inhaled Placebo
Drug: Inhaled Loxapine 5 mg — Inhaled Staccato Loxapine 5 mg, single dose
  Other Names: Inhaled Staccato Loxapine 5 mg; ADASUVE 5 mg
  Arms: Inhaled Loxapine 5 mg
Drug: Inhaled Loxapine 10 mg — Inhaled Staccato Loxapine 10 mg, single dose
  Other Names: Inhaled Staccato Loxapine 10 mg; ADASUVE 10 mg
  Arms: Inhaled Loxapine 10 mg

SUMMARY:
The purpose of this study is to assess efficacy and safety of Staccato Loxapine in the treatment of acute agitation in schizophrenic patients. The study will be conducted in 120 agitated schizophrenic patients - either newly admitted to a hospital setting or a research unit for acute agitation or already in hospital for chronic underlying conditions. Patients meeting entry criteria will be randomized to one of two doses of Staccato Loxapine or to Staccato Placebo. Following administration of study drug, assessment of agitation state will be conducted at serial time points using standard agitation scales over a 24 hour period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 to 65 years, inclusive.
2. Patients who have met DSM-IV criteria for schizophrenia, schizophreniform disorder, or schizoaffective disorder.
3. Patients who are judged to be clinically agitated at Baseline with a total score of ≥ 14 on the 5 items (poor impulse control, tension, hostility, uncooperativeness, and excitement) comprising the PANSS Excited Component (PEC).
4. Patients who have a value of ≥ 4 (out of 7) on at least 1 of the 5 items on the PANSS Excited Component.
5. Patients who read and understand English and provide written informed consent.
6. Patients who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, urinalysis and in the opinion of the Principal Investigator.
7. Female participants, if of child-bearing potential and sexually active, and male participants, if sexually active with a partner of child-bearing potential, who agree to use a medically acceptable and effective birth control method throughout the study and for one week following the end of the study. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm with spermicide, intrauterine device (IUD), condom with foam or spermicide, vaginal spermicidal suppository, surgical sterilization and progestin implant or injection. Prohibited methods include: the rhythm method, withdrawal, condoms alone, or diaphragm alone.

Exclusion Criteria:

1. Patients with agitation caused by acute intoxication must be excluded. Positive identification of non-prescription drugs during urine screening excludes the subject.
2. Patients treated with benzodiazepines or other hypnotics or oral or short-acting intramuscular antipsychotics within 4 hours prior to study drug administration must be excluded.
3. Patients treated with injectable depot neuroleptics within one dose interval prior to study drug administration must be excluded.
4. Patients with a history of allergic reactions to loxapine or amoxapine must be excluded.
5. Female patients who have a positive pregnancy test at screening or are breastfeeding must be excluded.
6. Patients who have Parkinson's disease, hydrocephalus, seizure disorder, or history of significant head trauma must be excluded.
7. Patients with laboratory or ECG abnormalities considered clinically significant by the investigator or qualified designee that would have clinical implications for the patient's participation in the study must be excluded.
8. Patients with serious and unstable illnesses including current hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease and congestive heart failure), endocrinologic, neurologic (including stroke, transient ischemic attack, subarachnoidal bleeding, brain tumor, encephalopathy, and meningitis), or hematologic disease must be excluded.
9. Patients who have a history of acute or chronic pulmonary disease that precludes administration of Staccato Loxapine (asthma, bronchitis, emphysema) must be excluded.
10. Patients who have received an investigational drug within 30 days prior to the current agitation episode must be excluded.
11. Patients who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving loxapine, or unable to use the inhalation device, must be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2006-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zimbroff, MD, Principal Investigator — Pacific Clinical Research Medical Group
Locations (1):
- Pacific Clinical Research Medical Group, 1317 West Foothill Blvd, Suite 200,, Upland, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Result] Allen MH, Feifel D, Lesem MD, Zimbroff DL, Ross R, Munzar P, Spyker DA, Cassella JV. Efficacy and safety of loxapine for inhalation in the treatment of agitation in patients with schizophrenia: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 Oct;72(10):1313-21. doi: 10.4088/JCP.10m06011yel. PMID 21294997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 centers between Sep-2006 and Jan-2007. Patients recruited for screening were: 1) admitted to a hospital or research unit with acute agitation, 2) inpatients being treated for chronic underlying conditions who presented with acute agitation, and 3) patients with agitation treated in a psychiatric ED.
Pre-assignment Details: Pre-Treatment Period was defined as the period immediately prior to dosing in which screening procedures and inclusion/exclusion criteria were used to evaluate all patients for eligibility to participate in the study.
Period: Overall Study
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Started | 43 | 45 | 41
Completed | 43 | 45 | 40
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg | Total
Number analyzed (Participants) | 43 | 45 | 41 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 45 | 41 | 129
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (7.7) | 40.8 (7.45) | 39.3 (8.77) | 41.2 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 7 | 24
  Male | 33 | 38 | 34 | 105
Region of Enrollment [Number; unit: participants]
  United States | 43 | 45 | 41 | 129

OUTCOME MEASURES:

1. Primary Outcome: PANSS-EC Change From Baseline
Description: The Positive and Negative Syndrome Scale-Excited Component (PANSS-EC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (min) to 7 (max). The PANSS-EC, the sum of these 5 subscales, thus ranges from 5 to 35. Individuals were eligible if they had a PANSS-EC of ≥14 (out of 35) and a score ≥4 (out of 7) on at least 1 of the 5 items.
Time Frame: 2 hours
Population: The ITT population consisted of all patients who took any study medication and had both baseline data and at least 1 efficacy assessment after the. Any observation recorded after the use of rescue medication was censored and subject to the last observation carried forward algorithm.
Measure: Mean (Standard Deviation); unit: PANSS units
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 43 | 45 | 41
PANSS units | -4.98 (4.13) | -6.71 (5.14) | -8.56 (4.9)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority; p = 0.0880, ANCOVA — p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p = 0.0002, ANCOVA — p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model

2. Secondary Outcome: BARS Change From Baseline After Drug Treatment
Description: Change from baseline on the Behavioral Activity Rating Scale (BARS) ranging from 1 to 7 where: 1 = difficult or unable to rouse, 2 = asleep but responds normally to verbal or physical contact, 3 = drowsy, appears sedated, 4 = quiet, and awake (normal level of activity), 5 = signs of overt (physical or verbal) activity, calms down with instructions, 6 = extremely or continuously active, not requiring restraint, 7 = violent, requires restraint.
Time Frame: 2 hours
Population: All patients receiving experimental treatment
Measure: Mean (Standard Deviation); unit: BARS Score, Change from Baseline, units
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 43 | 45 | 41
BARS Score, Change from Baseline, units | -0.930 (0.936) | -1.53 (1.38) | -2.02 (1.35)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority; p = 0.0583, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Clinical Global Impressions-Improvement Scale (CGI-I) After Drug Administration
Description: Clinical Global Impression- Improvement (CGI-I) scores ranged from 1 to 7: 0=not assessed (missing), 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: 2 hours
Population: All patients receiving treatment
Measure: Mean (Standard Deviation); unit: CGI-I Units (7=worse, 1=better)
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 43 | 45 | 40
CGI-I Units (7=worse, 1=better) | 3.19 (0.932) | 2.53 (1.10) | 2.28 (1.18)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority; p = 0.0067, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p = 0.0003, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: CGI-I Responders
Description: Frequency of response based on the CGI-I (defined as achieving a CGI-I score of 1 or 2 at 2 hours after administration of the inhalation)
Time Frame: 2 hours
Population: All patients treated
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 43 | 45 | 40
Participants | 9 | 22 | 25
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority; p = 0.0076, Fisher Exact
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p = 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: From informed consent through 30 days after last treatment
Description: Adverse events observed by the Investigator or study personnel during study assessments or when volunteered by the patient were recorded on the Adverse Event CRF. The severity of the AE and relationship to study drug was determined by the investigator. Medications used to treat the adverse event were recorded on the Concomitant Medication CRF.
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/45 | 1/41
Other Adverse Events (participants affected / at risk) | 14/43 | 14/45 | 16/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=43) | Inhaled Loxapine 5 mg (N=45) | Inhaled Loxapine 10 mg (N=41)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — A 43 year-old white male with a history of schizophrenia and intravenous drug abuse (heroin and cocaine) randomized to receive placebo, was found dead on the bathroom floor next to an empty syringe 6 days after treatment.
Worsening of hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — A 48 year-old m with schizophrenia on treatment for hypertension received Loxapine 5 mg. While being followed up as an out-patient (11 days later), he developed worsening hypertension (BP 210/130), was hospitalized, treated, and D/C the next day
Exacerbation of schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — A 23 year-old male with schizophrenia, randomized to receive Loxapine 10 mg, was hospitalized 14 days later for exacerbation of schizophrenia, agitation, noncompliance with medication taking and response to internal stimuli.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=43) | Inhaled Loxapine 5 mg (N=45) | Inhaled Loxapine 10 mg (N=41)
Dysgeusia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 7 (7)
Dizziness (Nervous system disorders) | 4 (4) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5)
Sedation (Nervous system disorders) | 6 (6) | 6 (6) | 9 (9)

LIMITATIONS AND CAVEATS:
Because of the need to provide informed consent, the types of patients enrolled in the study may not have been representative of the most severely agitated patients who present for emergency care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less